CLINICAL TRIAL: NCT00542256
Title: Effects of Transcranial DC Stimulation Coupled With Constraint Induced Movement Therapy on Motor Function in Stroke Patients
Brief Title: tDCS and Physical Therapy in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Study Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007P000420
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Cerebrovascular Accident
Keywords: Apoplexy; Cerebral Stroke; Cerebrovascular Accident, Acute; Cerebrovascular Apoplexy; Cerebrovascular Stroke; CVA (Cerebrovascular Accident); Stroke; Stroke, Acute; Vascular Accident, Brain
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): Each subject will receive 14 days (2 week period: 10 weekdays and 2 weekends) of constraint induced movement therapy. In addition, on the 10 weekdays during the treatment period, the subjects will come into the laboratory and receive up to 6 hours per day of training of the affected arm in a variety of tasks. At the beginning of each of the 10 weekday training sessions, participants will receive 40 minutes of active tDCS over the primary motor cortex.
  Interventions: Device: Active transcranial Direct Current Stimulation / Constraint Induced Movement Therapy
- 2 (Sham Comparator): Each subject will receive 14 days (2 week period: 10 weekdays and 2 weekends) of constraint induced movement therapy. In addition, on the 10 weekdays during the treatment period, the subjects will come into the laboratory and receive up to 6 hours per day of training of the affected arm in a variety of tasks. At the beginning of each training day tDCS will be applied for 40 minutes with the current active for only 30 seconds over the primary motor cortex.
  Interventions: Device: Sham transcranial Direct Current Stimulation / Constraint Induced Movement Therapy

INTERVENTIONS:
Device: Active transcranial Direct Current Stimulation / Constraint Induced Movement Therapy — 14 days of constraint induced movement therapy with 10 weekdays of up to 6 hours of training of the affected arm combined with application of tDCS over the primary motor cortex for 40 minutes.
  Arms: 1
Device: Sham transcranial Direct Current Stimulation / Constraint Induced Movement Therapy — 14 days of constraint induced movement therapy with 10 days of up to 6 hours of training in the affected arm and sham tDCS applied over the primary motor cortex for 40 minutes with active current applied for 30 seconds.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether a painless and noninvasive procedure called transcranial direct current stimulation (tDCS) combined with a method of physical therapy called constraint-induced movement therapy improves motor function in patients with chronic stroke. Research in healthy subjects has shown that when tDCS is combined with motor learning tasks, there is an increase in learning as compared to motor learning tasks only. The tDCS procedure sessions will be compared to sham (fake) procedure sessions, which is also called placebo stimulation. This study is double blind, which means neither the subjects nor researchers analyzing motor function will know if participants are receiving real tDCS stimulation or placebo. Only the person performing the procedure will know which one participants are receiving. Only by comparing the tDCS procedure to a sham (placebo) procedure can we understand if the tDCS actually improves motor function.

We hypothesize that tDCS will enhance the effects of constraint-induced movement therapy on motor recovery in chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* First time clinical ischemic or hemorrhagic cerebrovascular accident (radiologically confirmed)
* Demonstrates adequate balance while wearing a hand restraint on the unaffected arm
* Ability to stand from a sitting position and ability to stand with or without upper extremity support
* Stroke onset at least 6 months prior to study enrollment

Exclusion Criteria:

* Significant pre-stroke disability
* Any substantial decrease in alertness, language reception, or attention that might interfere with understanding instructions for motor testing
* Excessive pain in any joint of the paretic extremity
* A terminal medical diagnosis consistent with survival of less than 1 year
* Advanced liver, kidney, cardiac, or pulmonary disease
* Coexistent major neurological or psychiatric disease (including epilepsy)
* A history of significant alcohol or drug abuse in the prior 3 years
* Use of neuropsychotropic drugs - such as antidepressants
* Patients may not be actively enrolled in a separate intervention study targeting stroke recovery
* Patients may not have already received constraint-induced movement therapy and/or tDCS treatment for stroke

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-09; Primary Completion 2014-11-10 (Actual); Study Completion 2014-11-10 (Actual)

PRIMARY OUTCOMES:
Jebsen-Taylor Hand Function Test | Baseline, Treatment days 1,5,10, Follow Up
Motor Activity Log Rating Scale | Baseline, Treatment Days 1,5,10 and Follow Up
Beck Depression Inventory | Baseline, Treatment days 1,5,10 and Follow up
Visual Analogue Scale for Anxiety | Baseline, Treatment days 1,5,10 and Follow Up

SECONDARY OUTCOMES:
Fugl Meyer Assessment of Motor Recovery | Baseline Assessment
Barthel Index Score | Baseline Assessment
Modified Ashworth Scale | Baseline Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- See also: Related Info — http://www.tmslab.org